CLINICAL TRIAL: NCT00849290
Title: AN OPEN LABEL, SINGLE ARM TRIAL OF IMMUNOTHERAPY WITH AUTOLOGOUS ANTIGEN PRESENTING CELLS LOADED WITH PA2024 (APC8015F) FOR MEN WITH OBJECTIVE DISEASE PROGRESSION ON PROTOCOL D9902 PART B
Brief Title: Immunotherapy For Men With Objective Disease Progression On Protocol D9902 Part B (NCT00065442)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB01; NCT00090922 (obsolete NCT alias); NCT00170066 (obsolete NCT alias); NCT00513006 (obsolete NCT alias)
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Androgen Independent Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APC8015F (Experimental)
  Interventions: Biological: APC8015F

INTERVENTIONS:
Biological: APC8015F — APC8015F is an autologous active cellular immunotherapy product designed to stimulate an immune response against prostate cancer. APC8015F consists of autologous peripheral blood mononuclear cells (PBMCs), including antigen presenting cells (APCs), that have been activated in vitro with a recombinant fusion protein.

SUMMARY:
This is an open label, Phase 2 trial of APC8015F immunotherapy in men with objective disease progression on protocol D9902 part B (NCT00065442)

ELIGIBILITY:
Inclusion Criteria:

* Objective disease progression
* Subjects must have been enrolled in the APC-Placebo arm of D9902B (NCT00065442)

Exclusion Criteria:

* Infection requiring IV antibiotics
* Treatment with anticancer interventions within 14 days prior to enrollment
* Any medical condition which could compromise the study's objectives (discretion from sponsor)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Schellhammer, MD, Study Chair — Devine Tidewater Urology
Locations (58):
- United States (53):
  - UCLA, Los Angeles, California
  - USC Keck School of Medicine, Los Angeles, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Sharp HealthCare, San Diego, California
  - UCSF Cancer Center, San Francisco, California
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reid Army Medical Center, Washington D.C., District of Columbia
  - Miami Cancer Center, Miami, Florida
  - Hematology/Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Georgia Urology, P.A., Atlanta, Georgia
  - Midwest Prostate & Urology Health Center, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Lutheran General Cancer Center, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - Myron I Murdock MD LLC, Greenbelt, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic (Department of Urology), Burlington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Associates in Urology, LLC, West Orange, New Jersey
  - Albany Regional Cancer Center, Albany, New York
  - The Urological Institute of Northeastern New York, Albany, New York
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - New York Medical College, Hawthorne, New York
  - Beth Israel Cancer Center, New York, New York
  - Clinical Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - New York University, New York, New York
  - Staten Island Urological Research, Staten Island, New York
  - McKay Urology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - EACRI, Portland, Oregon
  - Kaiser Permanente Medical Group, Portland, Oregon
  - Center for Urologic Care, Bryn Mawr, Pennsylvania
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Mary Crowley, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Urology of Virginia, PC, Norfolk, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - University of Wisconsin, Madison, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - St. Luke's Hospital Immunotherapy Program, Milwaukee, Wisconsin
- Canada (5):
  - Can-Med Medical Research, Inc., Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Sunnybrook & Women's College HSC, Toronto, Ontario
  - Hospital Notre Dame du CHUM, Montreal, Quebec

REFERENCES:
- See also: (National Prostate Cancer Coalition) — http://www.pcacoalition.org
- See also: (USTOO International) — http://www.ustoo.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were registered between April 2004 and January 2009 across 52 clinical trial sites.
Pre-assignment Details: Participants who had objective disease progression on Dendreon's Phase 3 trial D9902B (NCT00065442)and who were determined to have received placebo were screened for evaluation of subject eligibility and performance of baseline tests/procedures.
Groups:
- APC8015F: APC8015F (cryopreserved autologous PBMCs, including APCs, that have been thawed and then activated in vitro with a recombinant fusion protein). Each dose contains a minimum of 3 X 10^6 CD54+ cells administered intravenously; treatment is 3 doses approximately 2 weeks apart.
Period: Overall Study
Arm/Group | APC8015F
Started | 113
Completed | 58
Not Completed | 55
Not completed — Adverse Event | 3
Not completed — Death | 14
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 5
Not completed — Disease Progression | 20

BASELINE CHARACTERISTICS:
Groups:
- APC8015F: Subjects receiving APC8015F
Arm/Group | APC8015F
Number analyzed (Participants) | 113
Age, Continuous [Mean (Full Range); unit: years] | 70.0 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 113

OUTCOME MEASURES:

1. Primary Outcome: Safety of APC8015F by Review of Reported Adverse Events
Description: All subjects who received at least one infusion of APC8015F (N = 109) were included in the safety analysis set and were followed for safety. Refer to Serious Adverse Events and Other Adverse Events.
Time Frame: periodically over 24 months
Population: All participants who received at least one infusion of APC8015F
Measure: Count of Participants; unit: Participants
Groups:
- APC8015F: Subjects receiving at least one infusion of APC8015F
Arm/Group | APC8015F
Number analyzed (Participants) | 109
Participants | 109

ADVERSE EVENTS:
Time Frame: 4 years, 9 months
Description: All subjects who received at least 1 infusion of APC8015F (N=109) were followed for safety.
  Total no. affected (32) = the number of subjects who experienced at least one serious adverse event (SAE). Subjects may have had > 1 SAE. Total no. of SAEs may exceed the no. affected. Subjects with <1 occurrence of the same event are counted only once.
Arm/Group | APC8015F
Serious Adverse Events (participants affected / at risk) | 32/109
Other Adverse Events (participants affected / at risk) | 101/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APC8015F (N=109)
Anaemia (Blood and lymphatic system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 2
Puncture site haemorrhage (General disorders) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Spinal cord compression (Nervous system disorders) | 7
Hydronephrosis (Renal and urinary disorders) | 2
Obstructive uropathy (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 4
Ureteric obstruction (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Poor venous access (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APC8015F (N=109)
Anaemia (Blood and lymphatic system disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 21
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 19
Asthenia (General disorders) | 8
Chills (General disorders) | 26
Fatigue (General disorders) | 29
Pain (General disorders) | 10
Pyrexia (General disorders) | 19
Urinary tract infection (Infections and infestations) | 7
Weight decreased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 28
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Dizziness (Nervous system disorders) | 11
Spinal cord compression (Nervous system disorders) | 8
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Hydronephrosis (Renal and urinary disorders) | 7
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6
HYPERTENSION (Vascular disorders) | 6
HYPOTENSION (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A provision provides for sponsor review up to 45 days with the right to request modification based on disclosure of confidential information; extendable by 60 days to file a patent application.